CLINICAL TRIAL: NCT03996824
Title: Study of Viral Transduction of Human Auditory Sensory Cells for the Development of Gene Therapy
Acronym: TREATGENE
Status: Recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-081
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — inner ear cells collected during surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AAV viral transduction: Collection of inner ear cells during a non-conservative surgical approach (translabyrinthine or transotic).
  Interventions: Other: Peroperative collect of inner ear cells

INTERVENTIONS:
Other: Peroperative collect of inner ear cells — After obtaining an informed consent during the preoperative medical visit, and if a non-conservative approach (translabyrinthine or transotic) is decided, the collect of inner ear cells will be performed during surgical approach.
  The sample will be collect in a sterile tube, and carried to the laboratory were it will be placed bon cell culture.

SUMMARY:
Gene therapy is a promising strategy to treat hearing loss and vestibular disorders, and Associated adenovirus (AAV) is shown as a good viral vector for inner ear therapy in animal models.

This study aims to study in vitro viral transduction of AAV in human inner ear cells, collected during non-conservative surgeries for vestibular schwannoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Operative indication for a non-conservative resection of vestibular schwannoma, decided by the surgeon in accordance with the patient
* Informed consent obtained
* Patients with a french social protection (AME excluded)

Exclusion Criteria:

* Intravestibular or intra-cochlear extension of the tumor
* Pregnant woman
* Patient with administrative control
* Medical contra-indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical resection of vestibular schwannoma.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2027-02-18 (Estimated); Study Completion 2027-02-18 (Estimated)

PRIMARY OUTCOMES:
AAV transduction in inner ear cells | 10 days
  The transduction will be measured with immunostaining techniques

CONTACTS AND LOCATIONS:
Overall Officials: Ghizlene Lahlou, Study Director — Institut Pasteur
Locations (2):
- France (2):
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
  - Hôpital Pitié-Salpétrière, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No